CLINICAL TRIAL: NCT01265264
Title: A Randomized, Double-Blind, Dose-Response Study of the Safety and Efficacy of Oral Ulodesine Added to Allopurinol in Subjects With Gout Who Have Not Adequately Responded to Allopurinol Monotherapy
Brief Title: Study to Evaluate sUA Lowering Activity, Safety and Efficacy of Oral Ulodesine Added to Allopurinol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCX4208-203
Record Dates: First submitted 2010-12-20; First posted 2010-12-23 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-10

CONDITIONS: Gout; Hyperuricemia; Arthritis; Joint Disease
Keywords: Gout; hyperuricemia; arthritis; joint diseases; allopurinol
MeSH Terms: conditions — Gout; Hyperuricemia; Arthritis; Joint Diseases | interventions — ulodesine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ulodesine Placebo + Allopurinol 300mg (Experimental): Oral dose administered daily for 84 days.
  Interventions: Drug: ulodesine; Drug: Placebo
- ulodesine 5mg + Allopurinol 300mg (Experimental): Oral dose administered daily for 84 days.
  Interventions: Drug: ulodesine; Drug: Placebo
- ulodesine 10mg + Allopurinol 300mg (Experimental): Oral dose administered daily for 84 days.
  Interventions: Drug: ulodesine; Drug: Placebo
- ulodesine 20mg + Allopurinol 300mg (Experimental): Oral dose administered daily for 84 days.
  Interventions: Drug: ulodesine; Drug: Placebo
- ulodesine 40mg + Allopurinol 300mg (Experimental): Oral dose administered daily for 84 days.
  Interventions: Drug: ulodesine; Drug: Placebo

INTERVENTIONS:
Drug: ulodesine — Oral dose administered daily for 84 days.
Drug: Placebo — Oral dose administered daily for 84 days.

SUMMARY:
The purpose of this study is to determine whether ulodesine and allopurinol combined for 12 weeks are effective in treating gout in patients who are not adequately responding to allopurinol alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 to < 70 years
* Baseline sUA ≥ 6.0 mg/dL after at least 2 weeks of treatment on a stable 300 mg dose of allopurinol
* Documented diagnosis of gout according to the American Rheumatism Association --Preliminary Criteria for the Diagnosis of Gout
* Be willing and able to take colchicine 0.6 mg per day or naproxen 220-250 mg twice daily as prophylaxis for gout flares and, if needed, a single daily dose of a proton pump inhibitor to prevent gastrointestinal discomfort
* Female participants must:

  * Be sexually abstinent
  * Be surgically sterile
  * Be postmenopausal or on stable contraception
* Male participants must:

  * Be sexually abstinent
  * Be > 1 year post-vasectomy
  * Using condoms with spermicide with partners meeting female requirements

Exclusion Criteria:

* Unable to tolerate 300 mg allopurinol
* Unable to tolerate both colchicine 0.6 mg per day and naproxen 220-250 mg twice daily
* Prior participation in a clinical study with BCX4208
* Gout flare during the Screening Period that is resolved for less than 2 weeks prior to first treatment with BCX4208 or placebo (exclusive of chronic synovitis/ arthritis)
* Unstable angina, symptomatic arrhythmia, signs or symptoms compatible with New York Heart Association Class III or Class IV heart failure, history of long QT syndrome, or QTc interval < 350 msec or > 475 msec
* Poorly controlled hypertension (SBP > 160 mmHg or DBP > 100 mmHG at Screening or Baseline)
* Moderate or severe renal impairment and/or calculated creatinine clearance of < 60 mL/min(Cockroft-Gault method)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values > 2.0 x ULN
* CD4+ cell counts by flow cytometry < 500 cells/mm3
* Hemoglobin < 10 g/dL or > 18 g/dL males or < 10 g/dL or > 17 g/dL females White blood cell count < 3.7 x 109/L or > 11 x 109/L
* Female subjects who are pregnant, breastfeeding, or planning a pregnancy within the next 4 months
* Positive serology for hepatitis B surface antigen or hepatitis C or HIV type 1
* Immunocompromised or on systemic immunosuppressive medications or antirheumatic drugs (including anakinra and adrenocorticotropic hormone)from Screening to Day 92
* Azathioprine or 6-mercaptopurine within 14 days of first dose of allopurinol Hydrochlorothiazide in doses > 50 mg per day from Screening to Day 92
* Use of herbal/dietary supplements Screening to Day 92
* Recipient of any live or attenuated vaccine within 6 weeks of Screening
* Uric acid-lowering drugs other than allopurinol from Screening to Day 92 Systemic corticosteroids within 4 weeks prior to Day 1 (this does not include pulmonary or nasal inhaler containing corticosteroids, ophthalmic corticosteroids, joint injections, or low potency topical steroids)
* Investigational drug within 30 days prior to signing the ICF for this study
* Clinically significant and relevant drug allergies
* Chronic or recurrent infections (≥ 3 infections at the same site within 12 months)
* Cancer within 12 months-Except non-melanomatous localized skin cancer or completely excised and cured carcinoma-in-situ of uterine cervix or subjects who were previously treated for prostate or breast cancer if they currently are stable and have not been on chemo therapy within the last year prior to screening.
* Alcohol or drug abuse within 12 months of signing the ICF, or current substance dependence or abuse
* Other medical conditions which, in the opinion of the PI, would jeopardize the safety of the study subject or impact the validity of the study results.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the dose response of ulodesine when combined with Allopurinol on sUA. | Day 85
  Level of serum uric acid levels be measured at Day 85 to evaluate in subjects with Gout.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Hollister, MD, PhD, Study Director — BioCryst Pharmaceuticals
Locations (54):
- United States (54):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Malvern, Arkansas
  - Anaheim, California
  - Burbank, California
  - Irvine, California
  - La Mesa, California
  - Los Angeles, California
  - Oceanside, California
  - Palm Springs, California
  - Paramount, California
  - Sacramento, California
  - San Jose, California
  - Walnut Creek, California
  - West Covina, California
  - DeLand, Florida
  - Edgewater, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Oldsmar, Florida
  - Sanford, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Meridian, Idaho
  - Gurnee, Illinois
  - Brownsburg, Indiana
  - Newton, Kansas
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Lansing, Michigan
  - Olive Branch, Mississippi
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Greer, South Carolina
  - Rapid City, South Dakota
  - Bristol, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Tacoma, Washington